CLINICAL TRIAL: NCT06232291
Title: Observation of Safety and Tolerability Within 1 Year of the Use of R-ketamine / Placebo in Drug-resistant Depression
Status: Completed | Type: Observational
Sponsor: Medical University of Gdansk (Other)
Collaborators: Perception Neuroscience (Industry)
Responsible Party: Sponsor
Other Study IDs: NKBBN/12/2023
Record Dates: First submitted 2024-01-22; First posted 2024-01-30 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Treatment-Resistant Depression; Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant; Depressive Disorder, Major

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
An observational-comparative study, without interfering with the treatment, based on an operationalized interview.

DETAILED DESCRIPTION:
Patients with treatment-resistant depression constitute a significant proportion (even 30%) of patients diagnosed with major depressive disorder (MDD. Since 2014, there have been reports of a potential antidepressant effect of the R-ketamine stereoisomer. At the UCK Department of Psychiatry, a phase 2 clinical trial (2a) has been conducted since 2022 with the use of R-ketamine in the form of an intravenous solution, administered by an infusion pump to patients with drug-resistant depression (sponsor Perception Neuroscience, Inc., protocol PCN-101-21, NCT05414422). The available data from studies indicate a potential treatment-transformative effect of the drug, but do not provide comprehensive information on the long-term effects of treatment in terms of effectiveness, tolerability, and safety of R-ketamine use. The study is cognitive and comparative study, without interfering with the diagnostics, treatment, and rehabilitation. It aims to collect effectiveness and safety observations within 12 months of participation in the PCN-101-21 study, at quarterly intervals (3, 6, 9, 12 months, +/- 4 weeks), with particular emphasis on exacerbations of the underlying disease, hospitalization, correction of psychotropic treatment or functional impairment requiring support from social security authorities. The study does not involve additional diagnostic, therapeutic or rehabilitation goals and is a retrospective analysis performed during a single visit.

ELIGIBILITY:
Inclusion Criteria:

Expressing informed consent to participate in the study and earlier participation in the PCN-101-21 study on site.

Exclusion Criteria:

Informed consent withdrawal.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients participating in the PCN-101-21 study from March 4, 2022, on site.
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2023-04-21 (Actual); Primary Completion 2024-05-24 (Actual); Study Completion 2024-05-24 (Actual)

PRIMARY OUTCOMES:
Safety record post IMP exposure. | Single psychometric assessment is performed along with a structured interview covering a period of 12 months after participation in the study.
  time to event and its nature: exacerbation of symptoms, hospitalization, change of treatment, functional disorders requiring social support.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Gdańsk, Gdansk, Poland

IPD SHARING:
Plan to Share IPD: Yes
data repository at site, available on request
Supporting Information: Study Protocol, ICF, CSR

REFERENCES:
- [Derived] Wlodarczyk A, Slupski J, Szarmach J, Cubala WJ. Single arketamine in treatment resistant depression: Presentation of 3 cases with regard to sick-leave duration. Asian J Psychiatr. 2024 Jun;96:104016. doi: 10.1016/j.ajp.2024.104016. Epub 2024 Mar 22. PMID 38554563